CLINICAL TRIAL: NCT06134024
Title: The Assessment of Effectiveness and Safety of Double Pigtail Plastic Stents During Endoscopic Transmural Drainage of Post-inflammatory Pancreatic and Peripancreatic Fluid Collections With Use of Lumen-apposing Metal Stents (LAMS).
Brief Title: The Role of Double Pigtail Plastic Stents During Endoscopic Transmural Drainage of Pancreatic Fluid Collections.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nicolaus Copernicus University (Other)
Responsible Party: Principal Investigator, Mateusz Jagielski, Professor, Nicolaus Copernicus University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DGGOS/MJ/2/2023
Record Dates: First submitted 2023-11-12; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Pancreatitis, Acute; Pancreatitis, Acute Necrotizing; Pancreatic Pseudocyst; Pancreatic Necrosis; Pancreatitis, Chronic
Keywords: gastrointestinal endoscopy; transmural drainage; lams; double pigtail plastic stents; endoscopic drainage
MeSH Terms: conditions — Pancreatitis; Pancreatitis, Acute Necrotizing; Pancreatic Pseudocyst; Pancreatitis, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LAMS with Double Pigtail Plastic Stents (Experimental): The group of participants with post-inflammatory pancreatic and peripancreatic fluid collections with double pigtail plastic stents introduced through the LAMS during endoscopic transmural drainage.
  Interventions: Procedure: Introduction of double pigtail plastic stents through the LAMS during endoscopic transmural drainage of post-inflammatory pancreatic and peripancreatic fluid collections
- LAMS without Double Pigtail Plastic Stents (Active Comparator): The group of participants with post-inflammatory pancreatic and peripancreatic fluid collections without double pigtail plastic stents introduced through the LAMS during endoscopic transmural drainage.
  Interventions: Procedure: Endoscopic transmural drainage of post-inflammatory pancreatic and peripancreatic fluid collections with use of LAMS only

INTERVENTIONS:
Procedure: Introduction of double pigtail plastic stents through the LAMS during endoscopic transmural drainage of post-inflammatory pancreatic and peripancreatic fluid collections — During endoscopic procedure of endoscopic transmural drainage of post-inflammatory pancreatic and peripancreatic fluid collections the operator introduces double pigtail plastic stents through the LAMS.
  Arms: LAMS with Double Pigtail Plastic Stents
Procedure: Endoscopic transmural drainage of post-inflammatory pancreatic and peripancreatic fluid collections with use of LAMS only — During endoscopic procedure of transmural drainage of post-inflammatory pancreatic and peripancreatic fluid collections the operator introduces transmurally the LAMS only, without the double pigtail plastic stents.
  Arms: LAMS without Double Pigtail Plastic Stents

SUMMARY:
The goal of this clinical trial is to learn about clinical usefulness of double pigtail plastic stents during endoscopic transmural drainage of post-inflammatory pancreatic and peripancreatic fluid collections with use of lumen-apposing metal stents (LAMS).

The main question it aims to answer is:

Does introduction of double pigtail plastic stents through the LAMS increases efficacy and safety of endoscopic transmural drainage of post-inflammatory pancreatic and peripancreatic fluid collections?

DETAILED DESCRIPTION:
Acute pancreatitis (AP) of moderate-to-severe clinical course is associated with a high risk of local complications and organ failure leading to increased mortality. Pancreatic and peripancreatic fluid collections (PPFCs) that can appear in the late phase of pancreatitis can take the form of pancreatic pseudocysts and walled-off pancreatic necrosis (WOPN). These types of PPFCs are the most common local complications of acute and chronic pancreatitis. For many years, the traditional treatment of post-inflammatory PPFCs in the late phase of pancreatitis relied on surgical methods. However, there has been a recent dynamic development of minimally invasive techniques, including endoscopic transluminal methods. While endoscopic treatment is an established method of managing these complications, some aspects of endotherapy are still a source of much controversy. One of the most debated issues in interventional endoscopy of local complications in pancreatitis is the use of transmural self-expanding metallic stents (SEMSs).

Endoscopic transmural drainage consists of creating a fistula between the lumen of the PPFC and gastrointestinal tract to allow for a free outflow of fluid out of the PPFC and into the gastrointestinal tract. During an endoscopic ultrasound (EUS)-guided procedure of endoscopic transmural drainage of post-inflammatory PPFCs, this can be visualized in the endosonographic image through the wall of the upper gastrointestinal tract. Afterwards, a transmural puncture of the PPFC is performed under EUS guidance and widened with a cystotome to a diameter of 10 Fr using coagulation. This forms a transmural cystostomy, which joins the gastrointestinal tract and the lumen of the PPFC. The next step of the endoscopic procedure is mechanical (with a dilator) or pneumatic (with a high-pressure balloon) dilation of the pancreaticocystogastrostomy or pancreaticocystoduodenostomy. Once dilated, a transmural SEMS or plastic stent(s) is introduced through the cystostomy to facilitate free passive transmural drainage of the collection contents into the gastrointestinal tract. Passive transmural drainage is an effective method of endoscopic treatment of pancreatic pseudocysts, whose contents are entirely liquid. In the case of necrotic PPFCs that contain both liquefied necrotic material and tissue fragments, it is necessary to use active transmural drainage, which consists of inserting an additional nasal drain through the transmural cystostomy to enable flushing of the collection cavity in the postoperative period.

The development of advanced endoscopic techniques has led to rapid advancements in biomedical materials, including polymers for manufacturing endoscopic devices. Currently, there is a wide variety of transmural endoprostheses of different sizes, shapes, and designs for endoscopic treatment of post-inflammatory PPFCs. These endoprostheses were divided into two groups. The first group includes plastic stents, usually made of Teflon or polyethylene. The second group is SEMSs, often referred to as "lumen-apposing metal stents" (LAMSs), that are used in the treatment of post-inflammatory pancreatic local complications. For many years, the only type of endoprosthesis available for use in transmural drainage was plastic double-pigtail stents. However, LAMSs have been attracting increasing interest as a relatively new option in endoscopy. LAMSs are a special type of SEMS used in a variety of gastrointestinal endoscopic procedures. They are made of nitinol wire and are fully covered with a silicone membrane.

However, the role of LAMSs in transmural drainage remains unclear. Many authors believe that use of LAMS during endoscopic transmural drainage increases risk of complications in form of bleeding. Despite the development of advanced endoscopic techniques and devices, the high rates of bleeding into the PPFC lumen remain a major challenge in transmural drainage treatment. This type of complication is often caused by blood vessels adjacent to the fluid collection being damaged by the distal flange of the LAMS. It seems that inserting a plastic double-pigtail stent through the LAMS limits the risk of this kind of complication by moving the back wall of the PPFC away from the distal flange, PPFC cavity bleeding during transmural drainage is still a major complication associated with a high risk of fatal outcomes.

In this trial the participants with post-inflammatory PPFCs will be divided into two arms.

The first arm will consist of participants who underwent traditional transmural drainage procedure with use of LAMS only.

The second arm will consist of participants with PPFCs who underwent endoscopic transmural drainage with use of LAMS and during the procedure double pigtail plastic stents will be introduced through the LAMS in order to prevent bleeding.

Each arm will consist of at least 50 participants with post-inflammatory PPFCs.

ELIGIBILITY:
Inclusion Criteria:

* participants of both sexes aged above 18 years
* participants, who provided informed consent for such treatment
* eligibility for transmural endoscopic drainage of post-inflammatory pancreatic and peripancreatic fluid collections procedure according to current medical knowledge based on evidence-based medicine.

Exclusion Criteria:

* pregnancy, breastfeeding, or intention to become pregnant during the study
* contraindications to electrosurgical instruments
* allergy to any of the materials used in the study
* participants ineligible for endoscopic treatment
* participants ineligible for general anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of efficacy of endoscopic transmural drainage of post-inflammatory pancreatic and peripancreatic fluid collections with use of double pigtail plastic stents introduced through the LAMS. | 12 months
  Evaluation of efficacy based on clinical picture and results of imaging examinations.
Rate of safety of endoscopic transmural drainage of post-inflammatory pancreatic and peripancreatic fluid collections with use of double pigtail plastic stents introduced through the LAMS. | 12 months
  Evaluation of safety based on clinical picture and results of imaging examinations.

SECONDARY OUTCOMES:
Rate of early complications during endoscopic transmural drainage of post-inflammatory pancreatic and peripancreatic fluid collections with use of double pigtail plastic stents introduced through the LAMS. | 30 days
  Evaluation of early complications within thirty days from onset of endoscopic drainage.
Rate of late complications during endoscopic transmural drainage of post-inflammatory pancreatic and peripancreatic fluid collections with use of double pigtail plastic stents introduced through the LAMS. | 12 months
  Evaluation of late complications of endoscopic drainage.
Rate of clinical success of endoscopic transmural drainage of post-inflammatory pancreatic and peripancreatic fluid collections with use of double pigtail plastic stents introduced through the LAMS. | 3 months
  Assessment of clinical results of endoscopic transmural drainage of post-inflammatory pancreatic and peripancreatic fluid collections with use of double pigtail plastic stents introduced through the LAMS.
Rate of long-term success of endoscopic transmural drainage of post-inflammatory pancreatic and peripancreatic fluid collections with use of double pigtail plastic stents introduced through the LAMS. | 24 months
  Assessment of long-term results of endoscopic transmural drainage of post-inflammatory pancreatic and peripancreatic fluid collections with use of double pigtail plastic stents introduced through the LAMS.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thoeni RF. The revised Atlanta classification of acute pancreatitis: its importance for the radiologist and its effect on treatment. Radiology. 2012 Mar;262(3):751-64. doi: 10.1148/radiol.11110947. PMID 22357880
- [Background] Sarr MG. 2012 revision of the Atlanta classification of acute pancreatitis. Pol Arch Med Wewn. 2013;123(3):118-24. doi: 10.20452/pamw.1627. Epub 2013 Jan 25. PMID 23396317
- [Background] Manrai M, Kochhar R, Gupta V, Yadav TD, Dhaka N, Kalra N, Sinha SK, Khandelwal N. Outcome of Acute Pancreatic and Peripancreatic Collections Occurring in Patients With Acute Pancreatitis. Ann Surg. 2018 Feb;267(2):357-363. doi: 10.1097/SLA.0000000000002065. PMID 27805963
- [Background] Freeman ML, Werner J, van Santvoort HC, Baron TH, Besselink MG, Windsor JA, Horvath KD, vanSonnenberg E, Bollen TL, Vege SS; International Multidisciplinary Panel of Speakers and Moderators. Interventions for necrotizing pancreatitis: summary of a multidisciplinary consensus conference. Pancreas. 2012 Nov;41(8):1176-94. doi: 10.1097/MPA.0b013e318269c660. PMID 23086243
- [Background] Arvanitakis M, Dumonceau JM, Albert J, Badaoui A, Bali MA, Barthet M, Besselink M, Deviere J, Oliveira Ferreira A, Gyokeres T, Hritz I, Hucl T, Milashka M, Papanikolaou IS, Poley JW, Seewald S, Vanbiervliet G, van Lienden K, van Santvoort H, Voermans R, Delhaye M, van Hooft J. Endoscopic management of acute necrotizing pancreatitis: European Society of Gastrointestinal Endoscopy (ESGE) evidence-based multidisciplinary guidelines. Endoscopy. 2018 May;50(5):524-546. doi: 10.1055/a-0588-5365. Epub 2018 Apr 9. PMID 29631305
- [Background] Baron TH, DiMaio CJ, Wang AY, Morgan KA. American Gastroenterological Association Clinical Practice Update: Management of Pancreatic Necrosis. Gastroenterology. 2020 Jan;158(1):67-75.e1. doi: 10.1053/j.gastro.2019.07.064. Epub 2019 Aug 31. PMID 31479658
- [Background] da Costa DW, Boerma D, van Santvoort HC, Horvath KD, Werner J, Carter CR, Bollen TL, Gooszen HG, Besselink MG, Bakker OJ. Staged multidisciplinary step-up management for necrotizing pancreatitis. Br J Surg. 2014 Jan;101(1):e65-79. doi: 10.1002/bjs.9346. Epub 2013 Nov 22. PMID 24272964
- [Background] Szeliga J, Jackowski M. Minimally invasive procedures in severe acute pancreatitis treatment - assessment of benefits and possibilities of use. Wideochir Inne Tech Maloinwazyjne. 2014 Jun;9(2):170-8. doi: 10.5114/wiitm.2014.41628. Epub 2014 Apr 1. PMID 25097683
- [Background] Bazerbachi F, Sawas T, Vargas EJ, Prokop LJ, Chari ST, Gleeson FC, Levy MJ, Martin J, Petersen BT, Pearson RK, Topazian MD, Vege SS, Abu Dayyeh BK. Metal stents versus plastic stents for the management of pancreatic walled-off necrosis: a systematic review and meta-analysis. Gastrointest Endosc. 2018 Jan;87(1):30-42.e15. doi: 10.1016/j.gie.2017.08.025. Epub 2017 Sep 1. PMID 28867073
- [Background] Beran A, Mohamed MFH, Abdelfattah T, Sarkis Y, Montrose J, Sayeh W, Musallam R, Jaber F, Elfert K, Montalvan-Sanchez E, Al-Haddad M. Lumen-Apposing Metal Stent With and Without Concurrent Double-Pigtail Plastic Stent for Pancreatic Fluid Collections: A Comparative Systematic Review and Meta-Analysis. Gastroenterology Res. 2023 Apr;16(2):59-67. doi: 10.14740/gr1601. Epub 2023 Apr 28. PMID 37187554
- [Background] Saumoy M, Kahaleh M. Superiority of metal stents for pancreatic walled-off necrosis: bigger is better! Gastrointest Endosc. 2017 Jun;85(6):1253-1254. doi: 10.1016/j.gie.2017.03.008. No abstract available. PMID 28522015
- [Background] Jagielski M, Smoczynski M, Szeliga J, Adrych K, Jackowski M. Various Endoscopic Techniques for Treatment of Consequences of Acute Necrotizing Pancreatitis: Practical Updates for the Endoscopist. J Clin Med. 2020 Jan 1;9(1):117. doi: 10.3390/jcm9010117. PMID 31906294